CLINICAL TRIAL: NCT03574961
Title: A Randomized Controlled Trial of e-Support in Persons With Multiple Sclerosis
Brief Title: E-Support Groups in Multiple Sclerosis
Acronym: eSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Victoria M. Leavitt, Assistant Professor of Neuropsychology (in Neurology and Gertrud, Dept of Neur Neuropsychology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR4052
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: depression; social isolation
MeSH Terms: conditions — Multiple Sclerosis; Depression; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Support Group (Experimental): Participants in this arm will receive the treatment, 12 weeks of 1-hr weekly moderated e-Support sessions.
  Interventions: Behavioral: e-Support group
- e-Journaling Placebo (Placebo Comparator): Participants in this arm will complete 12 weeks of 1-hr weekly online journaling activities.
  Interventions: Behavioral: e-Journaling placebo

INTERVENTIONS:
Behavioral: e-Support group — Online (remote), web-based support group via private video link.
  Other Names: e-Support
  Arms: e-Support Group
Behavioral: e-Journaling placebo — Online journaling activity.
  Other Names: e-Journaling
  Arms: e-Journaling Placebo

SUMMARY:
Primary objectives:

* To determine the feasibility of program (80% retained with 75% overall attendance, and completed immediate follow-up questionnaires from 75% of participants).
* To determine the efficacy of program (evaluated by decreased loneliness, operationalized as decreased total score on the UCLA Loneliness Scale from pre to post intervention).

Secondary objective:

* To determine whether program will affect depression and quality of life.

DETAILED DESCRIPTION:
This study involves prospective data collection from an intervention to investigate the impact of participation by MS patients in a 12-week guided online social support group. All outcomes will be compared to active control group. At the completion of a 12-week interval, all participants (placebo and treatment) will complete follow-up questionnaires. Three months after completing, participants will be sent follow-up questionnaires that will be evaluated as a 6-month follow-up, to assess retention of benefits.

Social support has been linked to better health outcomes in many clinical populations. Multiple sclerosis (MS), a chronic neurological disease that affects over 400,000 people in the United States, involves physical and cognitive disability that can have negative consequences on social integration. This can lead to social isolation, which may be dynamically related to depression, fatigue, and disease progression. The aim of the present study is to investigate the impact of support group involvement on persons with MS. Outcomes of interest include mood, loneliness, and quality of life (QOL). Many people with MS feel isolated and are unable to participate in support groups that meet in locations that may be far from home, difficult to travel to (due to physical disability or lack of resources), or may not be convenient for their schedules. Another hindrance is the apprehension that MS patients sometimes experience when they encounter patients with severe physical disability, or worse impairment than their own. For these reasons, the study is introducing remote support groups to be conducted via the internet, "e-Support." Attending a remote, internet based support group may be more appealing to patients with MS as it obviates the need to travel, thereby reducing cost, time, and energy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (any disease type)
* Age 18 or over
* Willingness to sign informed consent document

Exclusion Criteria:

* Unable to obtain access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of enrolled participants who completed follow-up questionnaires | 12 weeks
  Assess feasibility of the program: to retain and obtain completed questionnaires at immediate follow-up from 80% of enrolled participants (meeting the criteria of 75% attendance).
Change in UCLA Loneliness Scale total score (please note that the official name of the scale is the UCLA Loneliness Scale). | Baseline, 12 weeks (immediate follow-up)
  Assess efficacy of the program to decrease loneliness as defined by a significant decrease in total score on UCLA Loneliness Scale. This name never appears as anything other than UCLA Loneliness Scale, i.e. Russell 1996)

SECONDARY OUTCOMES:
Change in overall depression [Patient Health Questionnaire (PHQ-9)] total score | Baseline, 12 weeks
  Assess efficacy of the program to decrease depression as defined by a significant decrease in total score on Patient Health Questionnaire (PHQ-9): an efficient tool for depression screening. The scale ranges from 0-27, with higher scores indicating worse depression.
Change in overall Functional Assessment of Multiple Sclerosis Quality of Life (FAMS QoL) score | Baseline, 12 weeks
  Assess efficacy of the program to improve quality of life. The Functional Assessment of Multiple Sclerosis (FAMS) quality of life (QoL) instrument is a disease-specific, self-report questionnaire. It includes 7 subscales. The total score is generated by summing scores across all subscales, and ranges from 0-232, with higher scores reflective or worse overall function. In addition to considering a significant decrease in the total score as an indication of better overall function, we will separately examine each subscale to see whether decreases in score (indicating improvements in function) are shown. This includes the following subscales: mobility, symptoms, emotional well-being, general contentment, thinking and fatigue, family/social well-being, and additional concerns scales.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Leavitt, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center (MS Center), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided